CLINICAL TRIAL: NCT04389346
Title: A Cone Beam Computed Tomographic Evaluation of Healing of Apicomarginal Defects Using Autologous Platelet Aggregates : A Randomized Controlled Trial
Brief Title: A Cone Beam Computed Tomographic Evaluation of Healing of Apicomarginal Defects Using Autologous Platelet Aggregates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ankita Ramani
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-04

CONDITIONS: Chronic Apical Periodontitis
Keywords: Apicomarginal defects; Cone Beam Computed Tomography; Autologous platelet aggregate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with PRF group (Active Comparator): Autologous platelet aggregate (PRF) will be placed over the denuded root surface, following apicoectomy and before flap repositioning.
  Interventions: Procedure: Periapical surgery using autologous platelet aggregate
- Control group without PRF (Placebo Comparator): Flap will be repositioned following apicoectomy without placement of any autologous platelet aggregate.
  Interventions: Procedure: Periapical surgery without autologous platelet aggregate

INTERVENTIONS:
Procedure: Periapical surgery using autologous platelet aggregate — PRF will be placed over the denuded root surface, following apicoectomy and before flap repositioning
  Arms: Periapical surgery with PRF group
Procedure: Periapical surgery without autologous platelet aggregate — Flap will be repositioned following apicoectomy directly without placing any platelet aggregate
  Arms: Control group without PRF

SUMMARY:
This study will evaluate the effect of PRF (platelet rich fibrin) on the healing of apicomarginal defects. Healing of the defects will be assessed 2 dimensionaly by periapical radiograph and 3 dimensionaly using CBCT.

DETAILED DESCRIPTION:
Patients with apicomarginal defects as per the inclusion criteria will be randomly divided into two groups - (1) Test group - The denuded root surface will be covered by PRF (Choukron's method) and (2) Control group -No use of autologous platelet aggregate during periapical surgery. Radiographic and clinical healing will be assessed after 12 months, 2D healing will be assessed by Rud and Molven criteria and 3D healing will be assessed by Modified Penn 3D criteria.The clinical parameters recorded including periodontal pocket depth (PD), clinical attachment level (CAL) and gingival margin position (GMP) will be measured on buccal aspect of the interproximal space and mid buccal aspect of the involved teeth using Williams 'O' periodontal probe.Routine examination procedure will be used to evaluate any evidence of signs and/or symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A negative response to vitality tests with radiographic evidence of periapical radiolucency with no general medical contraindications for oral surgical procedures.
* Apicomarginal communication having probing depth > 6mm.
* Patients with no general medical contraindications for oral surgical procedures.
* Recurrent episodes of purulent discharge.
* Failed previous root canal treatment.
* Failed previous surgery with persistent bony lesion.
* Adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

* Clinical or radiographic evidence of root fracture.
* Resorptive processes involving more than apical third of the root.
* Any systemic disease contraindicating oral surgery including uncontrolled diabetes and pregnancy.
* Any condition effecting rate of healing like smoking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in periapical radiolucency | Baseline to 12 Months
  2 blinded caliberated operators will score the periapical radiolucency at baseline and 12 months by following scoring
  scores for 2D healing
  Score1-Complete healing defined by re-establishment of the lamina dura Score 2- Incomplete healing (scar tissue) Score 3- Uncertain healing Score 4- Unsatisfactory healing
  scores for 3D healing Score1- Complete healing Score 2- Limited healing Score 3- Uncertain healing Score 4- Unsatisfactory healing

SECONDARY OUTCOMES:
Clinical success | Baseline to 12 Months
  Clinical success will be assessed by absence of clinical signs and symptoms such as pain, swelling , sinus or tenderness on palpation or percussion

CONTACTS AND LOCATIONS:
Overall Officials: ANKITA RAMANI, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Ankita Ramani, Rohtak, Haryana, India